CLINICAL TRIAL: NCT05211687
Title: Smart Home-based Technology to Promote Functional Mobility Among Individuals With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Collaborators: Hebrew University of Jerusalem (Other); Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, Prinicipal Investigator, University of Haifa
Other Study IDs: GALITYS
Record Dates: First submitted 2022-01-02; First posted 2022-01-27 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
Keywords: parkinson's disease; Freezing of gait; Smart-home
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smart-home for freezing of gait — A projector, Kinect camera and computer are located 2 meters from the walking area. Participants walk nine times back and forth on the walking track, in each of three walking conditions:
  1. Baseline: participants walk in a comfortable pace. The walking track consist a rectangle created by a white light projected on the floor. Based on in this walking condition, step width and cadence are calculated to determine the individual parameters of the cueing.
  2. Light-stripes: The walking area consist of 4-5 white light-stripes. Space between the stripes is 110% of the participant step length. Participants are instructed to walk over the stripes.
  3. Metronome: The walking track consist of a rectangle created by a white light projected on the floor, and in addition metronome beats are delivered by the computer. Beats frequency are 90% of the cadence. Participants are instructed to match their steps to the metronome beats.
  Each walking condition up to 90 seconds.

SUMMARY:
Many patients with Parkinson's disease suffer of gait disorder termed as "freezing of gait" (FOG). non-pharmacological approach such as applying external cues is effective in mitigating FOG events. The aim of this study is to test the feasibility and patients satisfaction from a first stage of technology development, designed to deliver automatically external cues to the patients in their homes.

DETAILED DESCRIPTION:
People with Parkinson's disease (PwP) may experience severe difficulties in mobility that negatively affect their function and Quality of life. Freezing of gait, (FOG) is a brief and sudden inability to initiate walking or move forward, despite an intention to walk. Such episodes are often observed when PwP attempt to turn, cross a narrow space or negotiate obstacles. Rehabilitation interventions for FOG represent the most effective non-pharmacological approach to maintain functional independence and reduce the risk of falls. A key approach is the provision of external cues, defined as sensory stimuli, which facilitate gait initiation and continuation. These external cues are suggested to bypass the dysfunctional movement pathways in the basal ganglia and therefore, are considered effective in alleviating FOG. Cueing can be applied by different modalities; the most common are visual (e.g. spaced lines on the floor) and auditory (e.g. rhythmic metronome beats).

The term smart-home refers to a range of technologies that are designed for and deployed in individual residences, and are equipped with non-invasive, environmental, and physiological sensors. The concept of a "health smart-home" is a variation of smart-home with a focus on assistive technologies to enable the independence and wellness of residents, including the elderly and patients in supervised residences.

In this study, the investigators will be testing the first phase of developing a smart-home technology designed for patients coping with PD to use in their homes and aims to improve gait and assist in prevention of FOG. The aims of this exploratory study are to evaluate the 1) practical feasibility of the technology, 2) patient satisfaction and 3) the effect of the technology on gait. The device was developed by Selfit medical© and included application of light stripes (visual cues) and metronome beats (auditory cues) that are individually adjusted to the participant walking parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to walk independently
* The patient report on daily episodes of FOG as indicated by question #2 in the new FOG questionnaire ("How frequently do you experience freezing episodes?").
* Score>18 on the Telephone Version of the Mini-Mental State Examination (TMMSE)
* Intact hearing and vision by self-declaration

Exclusion criteria

• The patient suffer of any neurological condition other than Parkinson's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Poeple diagnosed with Parkinson's disease, living in the community
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of smart-home technology on step length (cm) | through study completion, an average of 1 year
  Step length (cm) is assessed during the three walking conditions in order to evaluate the effect of the cueing (visual and auditory) applied on gait.
  Data is collected by the Kinect sensor.
Effect of smart-home technology on step time (sec) are | Through study completion, an average of 1 year
  Step time (sec) is assessed during the three walking conditions in order to evaluate the effect of the cueing (visual and auditory) applied on gait.
  Data is collected by the Kinect sensor.
Feasibility and participants' satisfaction semi-structured interview | through study completion, an average of 1 year
  Following the walking session, participants answered questions in a semi-structured interview:
  1. Did you see the light stripes clearly? (Yes/no)
  2. Did you experience any discomfort while walking over the stripes? For example, did you feel dazzled?
  3. Did you feel any change in your walking while using the light stripes? (Yes/no)
  4. If you did feel any change, can you describe it in your own words?
  5. Try to evaluate the magnitude of change in walking using the following visual scale (ranging from -5 to 5 will be presented to the particpants, -5 represent "Much worse", 0 represent "No change" and 5 represent "Much better)
  6. Do you think that the light stripes would be effective for avoiding FOGs? Yes/No/ Maybe The same six questions are then asked about the metronome beats
  7. Would you like to have such technology installed at your home?
  8. If, yes, which kind of cues would you prefer (light stripe/ metronome)?
  9. Do you have any suggestion for improvement?

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yogev-Seligmann, PhD, Principal Investigator — University of Haifa
Locations (1):
- Galit Yogev-Seligmann, Haifa, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nieuwboer A, Rochester L, Herman T, Vandenberghe W, Emil GE, Thomaes T, Giladi N. Reliability of the new freezing of gait questionnaire: agreement between patients with Parkinson's disease and their carers. Gait Posture. 2009 Nov;30(4):459-63. doi: 10.1016/j.gaitpost.2009.07.108. Epub 2009 Aug 5. PMID 19660949
- [Background] Keus HSJ, Munneke M, G. M. et al. European Physiotherapy Guidline for Parkinson's Disease. (2014).
- [Derived] Yogev-Seligmann G, Josman N, Bitterman N, Rosenblum S, Naaman S, Gilboa Y. The development of a home-based technology to improve gait in people with Parkinson's disease: a feasibility study. Biomed Eng Online. 2023 Jan 19;22(1):2. doi: 10.1186/s12938-023-01066-2. PMID 36658571